CLINICAL TRIAL: NCT02830568
Title: Medical Economic Evaluation and of Quality of Life of the Kidney Living Donors. Comparison of the Taking of Kidney by cœliosurgery (Pure or " Hand-assisted "), by cœliosurgery Assisted by Robot and by the Classic Technique of Open Donor Nephrectomy.
Brief Title: Medical Economic Evaluation and of Quality of Life of the Kidney Living Donors.
Acronym: DOVIREIN
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 10.039
Record Dates: First submitted 2010-06-07; First posted 2016-07-13 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2010-05

CONDITIONS: Kidney Transplantation
Keywords: Kidney transplantation; Surgical procedures; Kidney living donors; Quality of life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- couples kidney living donor - receiver: Three groups for each technique of taking of kidney :
  1. open donor nephrectomy
  2. standard and hand-assisted laparoscopic donor nephrectomy
  3. laparoscopic robotic-assisted nephrectomy
  Interventions: Procedure: open donor nephrectomy; Procedure: standard and hand-assisted laparoscopic donor nephrectomy; Procedure: laparoscopic robotic-assisted nephrectomy

INTERVENTIONS:
Procedure: open donor nephrectomy — open donor nephrectomy
Procedure: standard and hand-assisted laparoscopic donor nephrectomy — standard and hand-assisted laparoscopic donor nephrectomy
Procedure: laparoscopic robotic-assisted nephrectomy — laparoscopic robotic-assisted nephrectomy

SUMMARY:
The main objective of this multicentre study is to conduct the evaluation of cost-efficiency of various techniques of kidney taking with regard the quality of life of the kidney living donors.

It will allow to compare three techniques of taking (open donor nephrectomy, cœliosurgery pure or " hand-assisted " and cœliosurgery assisted by robot) and to determine their respective advantages in quality of life, then their medico-economic consequences in a cost-efficiency approach from the point of view of the society.

The evaluation will concern the donor and the receiver followed three months after the taking.

The open donor nephrectomy will be the technique of reference with which will be compared the two others.

DETAILED DESCRIPTION:
Context : The most efficient treatment of the terminal chronic renal insufficiency is the renal transplantation, but in spite of the realization of more than 2000 transplants a year in France, the waiting list increases every year in a important way. The decrease of the offer of transplants from deathly donors led numerous countries to develop the renal transplant from alive donors. This type of transplantation represents in 2007 only 8,1 % of transplants in France (report of ABM on 2007), but the deficit in renal transplants and the new laws of bioethics should increase this donation (it represents until 70 % of the renal transplantations in certain centres of North America or the Northern Europe).

Although the French urology is at the top of the laparoscopic technique, the classic surgical taking by lombotomie stays the reference technique, practised by 58 % of the centres, with for the patient its consequences in terms of pain, of duration of hospitalization, convalescence and possible side effects. The development of the taking by cœliosurgery, mini-invasive technique, allowed to increase the number of wishes of organ donation in the centres which developed it. It is however a difficult technical gesture, requiring an important experience. This technique has the inconvenience of a more painful scar and more subject to complications than the section known pubic of "Pfannenstiel" used for the taking by pure cœliosurgery.

The surgical robot Da Vinci (Intuitive Surgical, Sunnyvale, California), with a 3D mink, the joints of the instruments inside the body, the reduction of the movements, the best ergonomics, improves the precision of the cœlioscopic gesture, but has a sharply upper cost. The CHU of Nancy was the pioneer in Europe to develop this technique from 2002, with very encouraging results on a series from now on more than 80 patients.

Only retrospective studies compared the quality of life between these techniques, and in spite of the major financial impacts (10 years of dialysis represent 100 K€; the price of the robot is of 1700 K€) and the important differences of quality of life according to these various surgical approaches, no prospective comparative medico-economic study was realized up to now. In France, where the hospital bears the load of all the expenses concerning the donor, including its daily allowances during its medical certificate, the shortening of the hospitalization and of the convalescence of the donor as well as the results improved by the transplantation at the receiver of a kidney living donor would allow a fast amortization of these expensive technologies.

Main objective : To compare the cost and the efficiency of the three techniques of taking of kidney living donor.

Main assessment criterion : The quality of life of the donor tested by generic measuring instruments EUROQOL and SF-36 (both to D-1 (the day before the renal transplantation), D4 (4 days after) and D90 (3 months after) and SF-36 to D-1 and D90). It will be realized at the donor's in preoperative (D-1), in postoperative (D4) and in the visit of follow-up in 3 months (D90). It will be also collected at the receiver's in preoperative (D-1), postoperative immediate (D4) and in the visit of follow-up in 3 months (D90).

The combination with the cost estimate will allow to build the marginal cost-efficiency ratio.

Secondary objectives envisaged:

* The evaluation of the quality of life of the receiver by measuring instrument becomes generic EUROQOL and SF-36 to D-1, D4 (only Euroqol) and D90.
* The comparison of the comfort of the surgeon and his physical and psychic investment by index card(form) of specific evaluation (Borg and NASA-TLX).
* The comparison of the coelio-surgical techniques : pure coelioscopy, coelioscopy " hand-assisted " and coelioscopy assisted by robot will concern the quality of life and the marginal cost-efficiency ratio.

ELIGIBILITY:
Inclusion Criteria:

* The receiver is registered on the ABM list;
* The receiver is on dialysis or in preterminal renal insufficiency;
* The donor is a member of the circle of acquaintances of the receiver.

Exclusion Criteria:

* Risk of difficulties of follow-up during 3 months following the transplant (ex: patient not living in France);
* Refusal of participation of the donor.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Couples living donor - receiver of the services of urology and nephrology of 24 CHU in France practicing one of three techniques :
  * Classic surgical taking by lombotomie : Besançon, Bicêtre, Caen, Lille, Marseille, Strasbourg, Tenon;
  * Taking by coeliosurgery pure or hand-assisted : Clermont-Ferrand, Créteil, Foch, Grenoble, La Pitié Salpêtrière, Lyon Sud, Montpellier, Nantes, Necker,Saint-Etienne,Saint-Louis,Toulouse, Rouen;
  * Coeliosurgical taking assisted by robot : Nancy, Nice, Lyon, Tours.
Sampling Method: Non-Probability Sample
Enrollment: 268 (Actual)
Dates: Start 2010-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Quality of life of the donor | D-1 (day before nephrectomy), D4 (4 days after nephrectomy) and D90 (90 days after nephrectomy)
  Quality of life of the donor as measured by EUROQOL (score 0 to 1) and SF 36 self-administered questionnaires (score 0 to 100 in each of 8 dimensions , at D-1 (the day before nephrectomy), D4 (4 days after nephrectomy) and D90 (90 days after nephrectomy).
  biological values of the donor and the receiver

SECONDARY OUTCOMES:
Sociodemographic data | D-1, the day before nephrectomy
  At D-1 (the day before nephrectomy), sociodemographic data are collected
Comfort, physical and mental investment of the surgeon measured by the Borg and the NASA-TLX scale | Day 0, the actual day of nephrectomy for each donor
  The Borg scale consists of 7 questions corresponding to the level of discomfort in 7 body segments of the surgeon with responses ranging from 0 (no discomfort) to 10 (very very strong discomfort). The surgeon is questioned every 30 minutes during the surgery. The NASA-TLX scale consists in 8 questions about physical and mental investment with responses ranging from 0 (low) to 100 (high). The surgeon completes this scale immediately at the end of the surgical procedure.
Biological values of the donor and the receiver | D-1 (day before nephrectomy), D2 (2 days after nephrectomy) D4 (4 days after nephrectomy) and D90 (90 days after nephrectomy)
  Blood count and serum electrolyte levels are collected. biological values of the donor and the receiver
Treatments administered to the donor | D0 (the actual day of nephrectomy for each donor), D2 (2 days after nephrectomy), D4 (4 days after nephrectomy) and D90 (90 days after nephrectomy)
  Treatments administered to the donor from D0 (the actual day of nephrectomy for each donor) to D90 (90 days after nephrectomy).
Medical exams performed on the donor | D-1 (day before nephrectomy), D2 (2 days after nephrectomy) D4 (4 days after nephrectomy) and D90 (90 days after nephrectomy)
  Medical exams performed on the donor from D0 (the actual day of nephrectomy for each donor) to D90 (90 days after nephrectomy).
Information on surgical technique employed to achieve nephrectomy and description of the graft. | Day 0, the actual day of nephrectomy for each donor
  Type of surgery (open donor nephrectomy, standard or hand-assisted laparoscopic donor nephrectomyor laparoscopic robotic-assisted nephrectomy), Duration of surgery and of ischemia and description of the graft.

CONTACTS AND LOCATIONS:
Locations (24):
- France (24):
  - CHU Saint Jacques de Besançon, Besançon
  - CHU Côte de Nacre de CAEN, Caen
  - CHU Montpied de Clermont-Ferrand, Clermont-Ferrand
  - CHU Henri Mondor, Créteil
  - CHU Hôpital Michallon de Grenoble, Grenoble
  - CHU Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Claude Huriez, Lille
  - CHU Lyon Sud, Lyon
  - Hôpital Edouard Herriot de Lyon, Lyon
  - CHU Hôpital de la Conception, Marseille
  - CHU Lapeyronie, Montpellier
  - CHU Brabois, Nancy
  - CHU Hôtel Dieu, Nantes
  - CHU Pasteur, Nice
  - Hôpital Necker, Paris
  - Hôpital Pitié Salpêtrière, Paris
  - Hôpital Saint-Louis, Paris
  - Hôpital Tenon, Paris
  - Hôpital Charles Nicolle, Rouen
  - CHU Saint Etienne, Saint-Etienne
  - CHU Hautepierre, Strasbourg
  - CMC Foch, Suresnes
  - Hôpital de Rangueil, Toulouse
  - CHU Bretonneau, Tours

REFERENCES:
- [Derived] Achit H, Guillemin F, Karam G, Ladriere M, Baumann C, Frimat L, Hosseini K, Hubert J. Cost-effectiveness of four living-donor nephrectomy techniques from a hospital perspective. Nephrol Dial Transplant. 2020 Nov 1;35(11):2004-2012. doi: 10.1093/ndt/gfz143. PMID 31377771